CLINICAL TRIAL: NCT02134756
Title: Impact of Nutritional Supplementation on Aerobic Performance and Fatigue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: USF-NS.Active-2014
Record Dates: First submitted 2014-04-11; First posted 2014-05-09 (Estimated); Results first posted 2020-12-07 (Actual); Last update posted 2020-12-07 (Actual); Status verified 2015-12

CONDITIONS: Performance; Fatigue
Keywords: Supplement impact; Performance; Fatigue
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- NutraStem Active (Experimental): Daily supplementation with NutraStem Active; 2 capsules per day for 28 days
  Interventions: Drug: NutraStem Active
- Placebo (Placebo Comparator): Daily supplementation with placebo; 2 capsules per day for 28 days
  Interventions: Drug: NutraStem Placebo

INTERVENTIONS:
Drug: NutraStem Active
  Arms: NutraStem Active
Drug: NutraStem Placebo
  Arms: Placebo

SUMMARY:
Compare an over-the-counter dietary supplement (NutraStem Active®) and placebo over a 30-day intervention on aerobic exercise performance and fatigue.

The hypothesis is that supplementation with NutraStem Active® improve aerobic performance and reduce subjective measures of fatigue.

DETAILED DESCRIPTION:
Compare an over-the-counter dietary supplement (NutraStem Active®) and placebo over a 30-day intervention on aerobic exercise performance and fatigue.

The hypothesis is that supplementation with NutraStem Active® improve aerobic performance and reduce subjective measures of fatigue.

The basic protocol includes baseline assessment of fitness and participation in a vigorous session of exercise immediately before and 30 days after consumption of the experimental supplement or placebo.

The exercise task is intended to be fatiguing and demanding but is not expected to create failure.

The supplement makes claims related to boosting exercise performance and reducing fatigue.

The study design will determine if these outcomes are in fact present in a group of healthy, young, and active adults.

The primary dependent measures are perceived exertion during exercise and levels of fatigue measured on multiple non-exercise days.

ELIGIBILITY:
Inclusion Criteria:

* healthy
* physically active
* non-smoker

Exclusion Criteria:

* known cardiovascular, pulmonary, or metabolic disease
* body mass index greater than 35

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2014-05; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marcus W Kilpatrick, PhD, Principal Investigator — University of South Florida; Danielle Williams, Study Director — University of South Florida
Locations (1):
- Health and Exercise Science Laboratory, Tampa, Florida, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- NutraStem Active; Placebo: 2 capsules per day for 28 days
Period: Overall Study
Arm/Group | NutraStem Active | Placebo
Started | 15 | 15
Completed | 14 | 13
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- NutraStem Active: Daily supplementation with NutraStem Active; 2 capsules per day for 28 days
  NutraStem Active
- Placebo: Daily supplementation with placebo; 2 capsules per day for 28 days
  NutraStem Active
- Total: Total of all reporting groups
Arm/Group | NutraStem Active | Placebo | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 15 | 30
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Perceived Exertion] | 23 (6) | 26 (7) | 25 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 14
  Male | 8 | 8 | 16
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30
Perceived Exertion [Mean (Standard Deviation); unit: units on a scale] | 7.5 (1.7) | 7.5 (1.8) | 7.5 (1.8)

OUTCOME MEASURES:

1. Primary Outcome: Perceived Exertion
Description: Ratings of perceived exertion (RPE) as measured on a self-report scale. The scale is a single-item measure ranging from 0 (no exertion) to 10 (max exertion).
Time Frame: 28 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NutraStem Active | Placebo
Number analyzed (Participants) | 14 | 13
units on a scale | 6.7 (2.0) | 7.4 (1.9)

2. Secondary Outcome: Perceived Fatigue
Description: Ratings of perceived fatigue as measured on a self-report scale. The scale is a single-item measure ranging from 1 (not at all) to 5 (extremely).
Time Frame: 28 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NutraStem Active | Placebo
Number analyzed (Participants) | 14 | 13
units on a scale | 5.8 (1.9) | 5.5 (2.4)

3. Secondary Outcome: Perceived Energy
Description: Ratings of perceived energy as measured on a self-report scale. The scale is a single-item measure ranging from 1 (not at all) to 5 (extremely).
Time Frame: 28 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NutraStem Active | Placebo
Number analyzed (Participants) | 14 | 13
units on a scale | 4.1 (1.7) | 4.6 (1.6)

ADVERSE EVENTS:
Arm/Group | NutraStem Active | Placebo
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No